CLINICAL TRIAL: NCT03484260
Title: Association Between the Prevalence of Cardiovascular Risk Factors and New Use of Testosterone
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19547
Record Dates: First submitted 2018-03-22; First posted 2018-03-30 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Hypogonadism
Keywords: Risk factors predicting the initiation of testosterone use
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Testosterone Product: Male subjects prescribed testosterone in UK
  Interventions: Drug: Testosterone Product
- Control group: Matched male subjects not prescribed testosterone in the UK

INTERVENTIONS:
Drug: Testosterone Product — Men used testosterone product following prescription
  Groups: Case group: Testosterone Product

SUMMARY:
We will investigate if testosterone is preferentially given to patients at higher risk of cardiovascular events. If this is the case, then observational studies may be prone to selection bias resulting in overestimation of the cardiovascular risk associated with testosterone when compared to a healthier population not taking testosterone

ELIGIBILITY:
Inclusion Criteria:

- All male individuals in the source population with a first testosterone use during the study period will be included as cases. The date of the GP consultation associated with the first testosterone prescription will be designated as the index day.

Exclusion Criteria:

- Patients of less than 18 years on the index day, with less than 2-year contribution to the CPRD-HES link before the index day, or with use of testosterone before the study period will be excluded from the group of cases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population is the subset of male patients in the Clinical Practice Research Datalink (CPRD) that has been linked to the Hospital Episodes Statistics (HES) database (CPRD-HES).
  Cases will be defined by first testosterone use between 1st January 2001 and 31st March 2016 (study period). The date of the GP consultation associated with the first testosterone prescription will be designated as the index day. All cases will be required to be over 18 years on the index day, to have contributed for at least 2 years to the CPRD-HES link and to have no history of testosterone before the index day.
Sampling Method: Non-Probability Sample
Enrollment: 27778 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Estimation of the association between cardiovascular risk factors and initiation of testosterone therapy | Retrospectively from 01 January 2001 to 31 March 2016

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Berlin, Germany